CLINICAL TRIAL: NCT03269552
Title: A Response-Adapted Clinical Trial of Weekly Carfilzomib With or Without Rituximab for Waldenström's Macroglobulinemia and Marginal Zone Lymphoma
Brief Title: Carfilzomib With or Without Rituximab in the Treatment of Waldenstrom Macroglobulinemia or Marginal Zone Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9702; NCI-2017-01548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9702 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1716046 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Marginal Zone Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory Marginal Zone Lymphoma; Refractory Waldenstrom Macroglobulinemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — carfilzomib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carfilzomib, rituximab) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who fail to achieve at least 25% M-protein reduction for Waldenstrom's macroglobulinemia or partial response for marginal zone lymphoma after 2 courses of carfilzomib, receive rituximab IV weekly on days 1, 8, 15, and 22 of course 3 and then monthly on day 1 of courses 4-6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This phase II trial studies how well carfilzomib with or without rituximab work in treating patients with Waldenstrom macroglobulinemia or marginal zone lymphoma that is previously untreated, has come back, or does not respond to treatment. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as rituximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving carfilzomib alone when disease is responding or with rituximab when disease is not responding may work better in treating patients with Waldenstrom macroglobulinemia or marginal zone lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate of single-agent weekly carfilzomib (CFZ), measured after 2 cycles of therapy, in Waldenstrom's macroglobulinemia (WM) and marginal zone lymphoma (MZL).

SECONDARY OBJECTIVES:

I. Assess safety and tolerability of single agent, weekly CFZ in patients with WM and MZL, and determine the tolerability of weekly CFZ+rituximab for applicable patients.

II. Estimate the time to best response, response duration, and survival with weekly CFZ for WM and MZL.

III. Evaluate the overall response rate associated with weekly CFZ in a subset of patients with rituximab refractory WM or MZL.

OUTLINE:

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who fail to achieve at least 25% M-protein reduction for Waldenstrom's macroglobulinemia or partial response for marginal zone lymphoma after 2 courses of carfilzomib, receive rituximab IV weekly on days 1, 8, 15, and 22 of course 3 and then monthly on day 1 of courses 4-6 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Waldenstrom's macroglobulinemia (WM) or marginal zone lymphoma (MZL) based on institutional pathology review; patients may have either previously untreated or relapsed/refractory disease
* Measurable disease: for WM presence of monoclonal IgM immunoglobulin concentration on serum electrophoresis, with lymphoplasmacytic marrow infiltrate; for MZL: measurable nodal disease measuring at least 1.5 cm in longest dimension, or splenomegaly
* Indication for initiation of therapy
* Absolute neutrophil count (ANC) > 1,000/uL unless disease-related (due to marrow infiltration or splenomegaly)
* Platelet count > 75,000/uL unless disease-related (due to marrow infiltration or splenomegaly)
* Serum creatinine < 2.5 mg/dL or creatinine clearance > 30 cc/min
* Bilirubin < 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Expected survival of > 90 days
* Females of childbearing potential (FCBP) must agree to pregnancy testing and to practice contraception
* Male subjects must agree to practice contraception

Exclusion Criteria:

* Known human immunodeficiency virus (HIV), hepatitis C, or hepatitis B positivity (subjects with hepatitis B surface antigen [SAg] or core antibody positivity, who are receiving and responding to antiviral therapy directed at hepatitis B or are negative for hepatitis B virus [HBV] deoxyribonucleic acid [DNA], are allowed)
* Candidate for potentially curative antibiotic therapy for gastric mucosa-associated lymphoid tissue (MALT); (gastric MALT lymphoma patients with stage I/II helicobacter [H.] pylori positive lymphoma must fail therapy with H.-pylori directed therapy before being considered for this study)
* Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher
* Known active central nervous system (CNS) involvement
* Pregnant or lactating females
* Inadequate cardiac function, as measured by left ventricular ejection fraction (LVEF) that is less than or equal to 40%, or the presence of New York Heart Association (NYHA) classification of greater than stage II congestive heart failure
* Significant neuropathy (grades 3-4, or grade 2 with pain) within 14 days prior to screening
* Uncontrolled inter-current illness including, but not limited to, unstable angina, recent myocardial infarction within 6 months of screening and uncontrolled cardiac arrhythmias, psychiatric illness, or psychosocial difficulty that would limit compliance with study requirements
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants signed informed consent, met eligibility and continued on to study treatment.
Groups:
- Treatment (Carfilzomib, Rituximab): Patients receive carfilzomib IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who fail to achieve at least 25% M-protein reduction for Waldenstrom's macroglobulinemia or partial response for marginal zone lymphoma after 2 courses of carfilzomib will continue to receive carfolzomib for 4 more courses. In addition, they will also receive rituximab IV weekly on days 1, 8, 15, and 22 of course 3 and then monthly on day 1 of courses 4-6 in the absence of disease progression or unacceptable toxicity.
  Carfilzomib: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Rituximab: Given IV
Period: Overall Study
Arm/Group | Treatment (Carfilzomib, Rituximab)
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Carfilzomib, Rituximab)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 64.25 [59 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Descriptive statistics will be used for baseline characteristics, and responses to treatment.
Time Frame: Up to 1 year
Population: Participants who were evaluated after cycle 2 day 15 and prior to cycle 3 day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carfilzomib, Rituximab)
Number analyzed (Participants) | 4
Participants
  Complete response | 0
  Very good partial response | 0
  Partial response | 2
  Minor response | 1
  Stable disease | 1
  Progressive disease | 0

2. Secondary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier analysis.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carfilzomib, Rituximab)
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Time to Best Response
Description: Estimated using Kaplan-Meier analysis.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Carfilzomib, Rituximab)
Number analyzed (Participants) | 3
Months | 2 [0.5 to 3]

4. Secondary Outcome: Time to Progression
Description: Estimated using Kaplan-Meier analysis.
Time Frame: Up to 1 year
Measure: Median (Standard Error); unit: Months
Arm/Group | Treatment (Carfilzomib, Rituximab)
Number analyzed (Participants) | 4
Months | 8 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the time the subject receives their first dose of study drug through 30 days post-last dose of study drug or initiation of a new anti-cancer therapy, whichever occurs first.
Arm/Group | Treatment (Carfilzomib, Rituximab)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carfilzomib, Rituximab) (N=4)
Microangiopathic Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carfilzomib, Rituximab) (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Cough (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Flatulance (Gastrointestinal disorders) | 2 (3)
Flu Like Symptoms (General disorders) | 1 (1)
Fluid Retention (General disorders) | 1 (1)
Warm Sensation (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Increased Cold Sensitivity (Nervous system disorders) | 1 (1) — In fingertips
Neutrophil Count Decreased (Investigations) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Platelet Count Decreased (Investigations) | 2 (3)
Decreased Urination (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
White Blood Cell Count Decreased (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to low accrual leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT03269552/Prot_SAP_000.pdf